CLINICAL TRIAL: NCT00824577
Title: Heart Rate Variability in Chronic Kidney Disease Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Jenq-Wen Huang, National Taiwan University Hospital
Other Study IDs: 200812010R
Record Dates: First submitted 2009-01-16; First posted 2009-01-19 (Estimated); Last update posted 2010-06-29 (Estimated); Status verified 2010-06

CONDITIONS: Chronic Kidney Disease; Heart Rate Variability
Keywords: heart rate variability; autonomic function; heart function
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — PD effluent and blood sample
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 250~300 patients: heart rate variability, heart function and Kt/V

SUMMARY:
Use 24hr Holter ECG, ultrasound and cardiac fibrosis markers in the chronic kidney disease patients

DETAILED DESCRIPTION:
24hr Holter examination is a non-invasive tool in detecting and diagnosing cardiac arrhythmia. Moreover, Heart rate variability has been proven to been an important prognostic factor in many cardiovascular diseases. The traditional linear analysis of heart rate variability proved to predict clinical outcome in myocardial infarction patients. The more delicate non-linear analysis in heart rate variability is one of the hot topics in the world.

Despite some biochemical values like WBC counts, platelet counts, BUN, creatinine, lactate, clinical vital parameters like blood pressure, heart rate, and oxygenation have been used to predict clinical outcome in chronic renal disease(CKD) patients, the application is still limited. It is an international interest to find a more safe and simple technique to identify important prognostic factors in CKD patients. Our project aimed to recruit these CKD patients from our hospital and conduct a cross-sectional study. Cardiac ultrasonography and 24hrs Holter will be arranged. Linear and non-linear analysis of heart rate variability will be performed and serum marker that influence prognosis like WBC count, platelet count, lactate, BUN, creatinine, fibrosis marker and adiponectin will be checked. Short term and long term outcome was followed and identify important prognostic factors to improve and detect clinical prognosis.

ELIGIBILITY:
Inclusion Criteria:

* peritoneal dialysis more than 3 months

Exclusion Criteria:

* pregnancy 2. received CT in recent 3 months

Ages: 15 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: peritoneal dialysis: peritoneal dialysis patient lasting for more than 3 months
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2009-12; Primary Completion 2010-06 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
heart rate variability, heart function, PET, Kt/V | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan